CLINICAL TRIAL: NCT04280380
Title: Incidence, Natural History and Outcome of Cytomegalovirus Infection in Critically Ill Patients and Patients Receiving Anticancer Therapy
Brief Title: Cytomegalovirus Infection in Critically Ill Patients and Patients Receiving Anticancer Therapy
Acronym: CMV-ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19.09.1441-GHM; HM-CMV19 (Other Grant/Funding Number: MSD)
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: CMV
Keywords: CMV; intensive care; prevalence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All eligible patients will be screened for CMV reactivation or primary infection until day 28 of ICU admission, discharge or death. For all eligible patients, a blood sample will be drawn for CMV serology and PCR testing at ICU admission (day 0) and then once a week for PCR testing (every Monday for logistic reasons) until day 28th of ICU admission, ICU discharge or death.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanical ventilated patients without cancer: This observational, cohort, retrospective and multicenter study will be performed during a period of 16 months at the 5 medical/surgical ICUs from HM Hospitals group.
  The recruitment will be performed by volume of patients: recruitment of the first 300 patients without cancer will start the 15th of January 2018 and will end once the last patient has been included; likewise, recruitment of the first patient with cancer will start on the same date and will end once the last patient (of 100) is recruited. Patients undergoing any type of anticancer therapy within the previous 3 month of ICU admission will be analyzed as part of the overall group but also as an independent subgroup of patients.
  Inclusion criteria: (a) age >=18 y.o., (b) admission to the intensive care unit with an expectancy to stay longer than 72 hours and requiring invasive mechanical ventilation.
  Interventions: Diagnostic Test: Real time PCR
- Mechanical ventilated patients with cancer: This observational, cohort, retrospective and multicenter study will be performed during a period of 16 months at the 5 medical/surgical ICUs from HM Hospitals group.
  The recruitment will be performed by volume of patients: recruitment of the first 300 patients without cancer will start the 15th of January 2018 and will end once the last patient has been included; likewise, recruitment of the first patient with cancer will start on the same date and will end once the last patient (of 100) is recruited. Patients undergoing any type of anticancer therapy within the previous 3 month of ICU admission will be analyzed as part of the overall group but also as an independent subgroup of patients.
  Inclusion criteria: (a) age >=18 y.o., (b) admission to the intensive care unit with an expectancy to stay longer than 72 hours and requiring invasive mechanical ventilation.
  Interventions: Diagnostic Test: Real time PCR

INTERVENTIONS:
Diagnostic Test: Real time PCR — At inclusion, serum samples will be collected to determine CMV serological status. Plasma samples will be collected weekly for CMV PCR analysis. Antibodies for CMV will be assessed using a commercial enzyme immunoassay kit for detection of total antibodies to CMV (LIAISON CMV IgG assay, DiaSorin S.p.A). DNA will be extracted in 200 μL of plasma eluted in 60 μL of elution buffer using a NucliSENS easyMAG system (bioMérieux, Boxtel, The Netherlands). Samples will be amplified using Affigene CMV Trender diagnostic assay (Cepheid AB, Bromma, Sweden), according to the manufacturer instructions. Amplification will be performed on a MX3000P instrument (Stratagene Instruments Systems, La Jolla, CA, USA). Samples with >500 copies/mL of plasma will be considered positive.

SUMMARY:
Cytomegalovirus (CMV) is the most common member of the herpes viruses to infect humans. Its double-stranded linear DNA duplex contains 165 genes that encode viral proteins that mimic and interact with human cellular proteins and are related to its virulence and latency. CMV primary infection is usually acquired in the adolescence and follows a benign course; however it might reactivate in patients with immune suppression leading to a high mortality and morbidity in this group of patients. There is growing evidence that critically ill immunocompetent patients can develop CMV disease [Limaye et al. JAMA. 2008;300(4):413; Ziemann et al. Crit Care Med. 2008;36(12):3145]. However, results of the incidence of CMV disease in critically ill patients is unpredictable due to the wide range of these results, from a 0% to 98% [Al-Omari et al. Ann. Intensive Care (2016) 6:110]. This inconsistency could be explained by many factors such as (i) variation in the definition of CMV disease (old studies consider seropositivity as evidence of disease, while others use newer technologies like PCR and/or antigen detection), (ii) variation in inclusion criteria (some studies include only seropositive patients therefore assessing reactivation rate of CMV, others also include seronegative patients thus evaluating also new infections) or (iii) variation in studied populations (e.g. septic, surgical, burn or postcardiac surgery patients or patients under mechanical ventilation).

DETAILED DESCRIPTION:
Evidence in the literature has demonstrated how different factors have been associated with CMV disease; however, the effect of new anticancer therapies (personalized chemotherapies, biological and immunological treatments, extreme surgery, etc.) on CMV disease is unknown. The investigators believe that studying this subgroup of patients should be one of the primary issues as the number of patients with these characteristics will increase significantly in the near future.

Likewise, it is important to point out that in the real world diagnosing CMV disease is a real challenge for the intensive care physician (due to subclinical or not specific clinical presentations, confusion factors, low clinical suspicions, etc.) thus its diagnosis and eventual treatment could be improved. These undesired diagnostic and therapeutic flaws provide a unique opportunity to (i) describe the natural evolution of the disease, (ii) address the effect of the disease in the outcome of the patients and (iii) estimate the potential number of patients that could benefit from a new management.

HM Hospitales (https://www.hmhospitales.com/) is a Spanish private group made up of five tertiary university hospitals in Madrid (HM Madrid, HM Torrelodones, HM Sanchinarro, HM Puerta del Sur y HM Monteprincipe). In addition, the group has a specialized center focused in cancer ("Clara Campal" oncologic center https://www.hmciocc.com/ ) with a phase I Unit (STAR-CIOCC http://startmadrid.com/index.php/en/2014-10-02-23-29-01/madrid-locations/2014-10-10-00-46-42), five medical-surgical ICUs (one in each hospital) that assist 1200 patients/year (35% with cancer) and a surgical department specialized in robotic and laparoscopic procedures.

To define the incidence of CMV reactivation and disease is of paramount importance as several studies have suggested an association between CMV disease and an increased mortality rate, prolonged mechanical ventilation as well as length of ICU and hospital stay. Furthermore, CMV disease increases the risk of acquiring a nosocomial infection that could also have an effect on the outcome of the patients [Ziemann et al. Crit Care Med. 2008;36(12):3145; Sinclair. J Clin Virol. 2008;41(3):180]. Likewise, as several anti-CMV treatments are (valacyclovir, valanciclovir, ganciclovir, foscarnet or cidofovir), or will be shortly (letermovir), available the increased morbidity and mortality associated to this infection in critically ill patients could be improved dramatically.

This research proposal is seeking to answer four questions in a general ICU cohort of patients and in the subgroup of critically ill patients receiving anti-cancer therapy:

1. Which is the incidence of CMV infection and disease?
2. What is the natural evolution of CMV infections that do not receive anti-CMV treatment?
3. What is the impact of anti-CMV treatment in the patient´s outcome (mortality, days under mechanical ventilation and days at ICU)?
4. What are the risk and protective factors for developing CMV infection after ICU admission?

ELIGIBILITY:
Inclusion Criteria:

1. age >=18 y.o.,
2. admission to the intensive care unit with an expectancy to stay longer than 72 hours and requiring invasive mechanical ventilation.

Exclusion Criteria:

1. survival expectation previous to ICU admission less than 6 months,
2. intubation after 12 hours of ICU admission
3. limitation of the therapeutic effort previous or during the ICU stay,
4. admission to the ICU during the previous 3 months
5. not agreeing to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with >=18 years old, after admission to the intensive care unit with an expectancy to stay longer than 72 hours and requiring invasive mechanical ventilation, whom are not included at exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytomegalovirus Prevalence | From study start date (March, 2020) until ending enrollment period (16 months later)
  Cytomegalovirus prevalence after admission to the intensive care unit with an expectancy to stay longer than 72 hours

IPD SHARING:
Plan to Share IPD: No
Scientific congress and JCR publications